CLINICAL TRIAL: NCT01545011
Title: Effects of Inspiratory Muscle Training Combined With a Pulmonary Rehabilitation Program Versus a Program of Pulmonary Rehabilitation Alone on Dyspnea: a Randomized Trial
Brief Title: Effects of Inspiratory Muscle Training on Dyspnea in Subjects With Chronic Obstructive Pulmonary Disease
Acronym: IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RB 11.083 (EMI)
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2012-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Inspiratory muscle training; COPD; Conventional respiratory rehabilitation; Dyspnea scale
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard (No Intervention): conventional respiratory rehabilitation
- IMT (Experimental): Inspiratory muscle training and conventional respiratory rehabilitation
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — Inspiratory muscle training
  Arms: IMT

SUMMARY:
The purpose of this study is to determinate whether inspiratory muscle training (IMT) associated with a conventional respiratory rehabilitation program is more effective than a conventional respiratory rehabilitation program alone,on Dyspnea in chronic obstructive pulmonary disease (COPD) subjects with a normal maximum inspiratory pressure (IP > 60 cmH2O).

DETAILED DESCRIPTION:
Dyspnea is the main complaint of patients with COPD. Dyspnea is explained largely by the distension, objectified by measuring inspiratory capacity (IC), which places the diaphragm at a disadvantage to be effective, which raises the sensation of dyspnea.

Currently, inspiratory muscles training is recommended by the French-language Society of Pneumology, in case of an objective reduction of the strength of these muscles (corresponding to maximum inspiratory pressure <60 cm H20).

ELIGIBILITY:
Inclusion Criteria:

* Patient with COPD
* Hospitalized in the pulmonary rehabilitation unit in the hospital of Morlaix, with a 3 weeks pulmonary rehabilitation course

Exclusion Criteria:

* Pneumonectomy, Lobectomy less than 6 months
* Cardio-pulmonary anomaly
* Max inspiratory pressure < 60 cm H2O

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Dyspnea measure | 21 days
  Measure of changes in Mutidimentionnal Dyspnea Profile result questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Brest University Hospital, Brest, Brittany Region
  - Hospital of Morlaix, Morlaix, Brittany Region

REFERENCES:
- [Result] Beaumont M, Mialon P, Le Ber-Moy C, Lochon C, Peran L, Pichon R, Gut-Gobert C, Leroyer C, Morelot-Panzini C, Couturaud F. Inspiratory muscle training during pulmonary rehabilitation in chronic obstructive pulmonary disease: A randomized trial. Chron Respir Dis. 2015 Nov;12(4):305-12. doi: 10.1177/1479972315594625. Epub 2015 Jul 13. PMID 26170421